CLINICAL TRIAL: NCT01256892
Title: Insulin Dependent Gestational Diabetes Mellitus: Randomized Trial of Induction of Labour at 38 and 40 Weeks of Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof.Dr. Peter Husslein
Other Study IDs: 244/2002
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Labor, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: induction of labour

SUMMARY:
To evaluate the impact of induction of labour at 38 weeks with the induction of labour at 40 weeks in women with insulin dependent gestational diabetes mellitus on maternal and fetal outcome.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with insulin dependent gestational diabetes mellitus

Exclusion Criteria:

* chronic inflammatory disease,
* autoimmune disease,
* pre-existing diabetes mellitus,
* previous cesarean section,
* multiple pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult